CLINICAL TRIAL: NCT05579938
Title: A Randomised, Double-blind Clinical Trial to Determine the Effect of a Lozenge Containing Enzymes on Dental Biofilm Accumulation in Healthy Adults Using a 4-day Plaque Regrowth Model.
Brief Title: Effect of Enzymes on Dental Biofilm Accumulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novozymes A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-NZ-03
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Dental Plaque
Keywords: Enzymes; Dental biofilm; Dental plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum Lozenges (Active Comparator): Active enzyme-containing lozenges to be consumed 5 times per day for 4 days
  Interventions: Dietary Supplement: Enzyme-containing lozenge
- Identical Placebo Lozenges (Placebo Comparator): Placebo lozenges to be consumed 5 times per day for 4 days
  Interventions: Dietary Supplement: Placebo lozenge

INTERVENTIONS:
Dietary Supplement: Enzyme-containing lozenge — A lozenge containing 3 active enzymes
  Arms: Verum Lozenges
Dietary Supplement: Placebo lozenge — Identical placebo lozenge
  Arms: Identical Placebo Lozenges

SUMMARY:
Double-blind, placebo-controlled, cross-over study investigating dental biofilm accumulation after 4-days in 28 subjects randomised to receive:

Sequence 1: 5 active enzyme-containing lozenges per day for 4-days followed by a 2-week washout period followed by 5 identical placebo lozenges per day for 4-days or

Sequence 2: 5 placebo lozenges per day for 4-days followed by a 2-week washout period followed by 5 identical active enzyme lozenges per day for 4-days

DETAILED DESCRIPTION:
28 healthy subjects (aged 18-75y) will be randomised to receive Sequence 1 or Sequence 2 in a double-blind, placebo-controlled cross-over study. Subjects will refrain from all mechanical oral hygiene over the course of each 4-day intervention period (e.g. no brushing, flossing, chewing gum) and will brush twice daily with a standard ADA accepted toothbrush and fluoride toothpaste during the 2-week washout period.

Sequence 1: 5 active enzyme-containing lozenges per day for 4-days followed by a 2-week washout period followed by 5 id entical placebo lozenges per day for 4-days or

Sequence 2: 5 placebo lozenges per day for 4-days followed by a 2-week washout period followed by 5 identical active enzyme lozenges per day for 4-days.

The primary outcome measure is 4-day biofilm accumulation as assessed by the Lobene-Soparkar Modification of the Turesky Modification of the Quigley-Hein Plaque Index score from Baseline (following dental prophy and score of 0) to Day 4 in the absence of oral mechanical hygiene (e.g. brushing, flossing).

The secondary outcome measure is 24-hour biofilm accumulation as assessed by the Lobene-Soparkar Modification of the Turesky Modification of the Quigley-Hein Plaque Index score from Baseline (following dental prophy and score of 0) to Day 1 (approximately 24-hours) in the absence of oral mechanical hygiene (e.g. brushing, flossing).

Exploratory measures include:

1. Shift in S. mutans relative abundance and richness (number of species) from baseline to Day 4 based on Next Generation Sequencing (alpha/beta diversity and individual Amplicon Sequence Variants [ASV] measured by 16S sequencing)
2. Shift in detected oral bacterial species of interest from baseline to Day 4, based on Next Generation Sequencing (alpha/beta diversity and individual Amplicon Sequence Variants [ASV] measured by 16S sequencing)
3. Change in IL-1-beta, IL-6, IL-8 and TNF-alpha from baseline to Day 4, based on electrochemiluminescence assay
4. Post-product use questionnaire (developed by sponsor) after 4 days of product use

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy males and females 18-75 years of age.
2. Able to read, sign and receive a copy of the signed informed consent form.
3. Have at least 20 natural teeth with scorable facial and lingual surfaces. A scorable tooth is defined as having at least 2/3 of the natural tooth surface evaluable for the selected clinical measurements. The following will not be included in the scorable tooth count: third molars; teeth that are fully crowned/extensively restored, grossly carious, orthodontically banded/bonded or abutment teeth; teeth exhibiting general cervical abrasion and/or enamel abrasion and calculus deposits which, in the opinion of the clinical examiner, would interfere with the assessments)..
4. Willing to refrain from all oral hygiene 8-12 hours prior to Screening visit.
5. Willing to refrain from use of chewing gum over the course of the 4-day intervention periods
6. At the Screening Visit, subject presents with:

   a. A plaque index score ≥ 1.95 according to the Lobene-Soparkar Modification of the Turesky Modification of the Quigley-Hein Plaque Index, following 8 to 12 hours plaque accumulation period.
7. Willing and able to comply with scheduled visits, treatment plan and other study procedures.
8. Willing to refrain from all oral hygiene (with the exception of lozenge consumption 5 times per day) for a 96-hour (4-day) period between Visits 2-4/Visits 5-7
9. Willing to refrain from the use of chemotherapeutic antiplaque/antigingivitis products containing antibacterial agents such as, but not limited to, amine fluoride, chlorhexidine, stannous fluoride, essential oils, cetylpyridinium chloride, etc. and other oral hygiene products during the study.

Exclusion Criteria:

1. A subject with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the subject inappropriate for entry into this study.
2. Subject self-reported as currently pregnant, or breastfeeding or subject intends to become pregnant through the duration of the study.
3. Uncontrolled diabetes or hypertension.
4. Health condition requirement for antibiotic premedication prior to dental procedures.
5. Current history of antibiotic, anti-inflammatory, anti-coagulant medication or chemotherapeutic antiplaque/antigingivitis therapy within 30 days of Screening visit.
6. Subject is a smoker or user of smokeless tobacco, nicotine containing products (including chewing gum, patches, pouches or mints).
7. Subject has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
8. Presence of moderate or severe periodontal disease (Stage II, III or IV), or actively under treatment for periodontal disease.
9. Presence of orthodontic appliances, peri/oral piercings, or removable partial dentures.
10. History of allergy or significant adverse events following use of oral hygiene products such as toothpastes, mouth rinses, breath mints, lozenges, or chewing gum or their ingredients.
11. A subject with high levels of extrinsic stain, calculus deposits or severely inflamed tissues which might interfere with dental plaque assessments.
12. Have significant intra-oral soft tissue lesions due to pathology or trauma based on a visual examination.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
4-day biofilm accumulation in the absence of oral mechanical hygiene | 4-day biofilm accumulation from Baseline following dental prophylaxis (score of 0) to Day 4
  Biofilm accumulation is assessed by the Lobene-Soparkar Modification of the Turesky Modification of the Quigley-Hein Plaque Index (PLI)

SECONDARY OUTCOMES:
24-hour biofilm accumulation in the absence of oral mechanical hygiene | 24-hour biofilm accumulation from Baseline following dental prophylaxis (score of 0) to 24-hours
  Biofilm accumulation is assessed by the Lobene-Soparkar Modification of the Turesky Modification of the Quigley-Hein Plaque Index (PLI)

OTHER OUTCOMES:
Abundance of salivary and plaque S. mutans | 4-days (Baseline to Day 4) for each crossover period
  alpha/beta diversity measured by 16S rRNA sequencing
Shift in detected plaque and saliva bacterial species of interest | 4-days (Baseline to Day 4) for each crossover period
  Analysis will be based on Next Generation Sequencing (alpha/beta diversity and individual Amplicon Sequence Variants [ASV] measured by 16S rRNA sequencing
Change in inflammatory markers from Baseline to Day 4 | 4-days (Baseline to Day 4)
  Analysis of IL-1-beta, IL-6, IL-8 and TNF-alpha will be based on electrochemiluminescence assay
Post-product use questionnaire | 4-days (Baseline to Day 4) for each crossover period
  Consumer-based questionnaire developed by Sponsor

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L Milleman, DDS, MPA, Principal Investigator — Salus Research Inc
Locations (1):
- Salus Research Inc, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No